CLINICAL TRIAL: NCT05206435
Title: Methadone-Maintained Smokers Switching to E-Cigarettes
Acronym: SHINE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1702236; R01DA052907 (NIH)
Record Dates: First submitted 2021-12-21; First posted 2022-01-25 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Nicotine Dependence; Electronic Cigarette Use
MeSH Terms: conditions — Tobacco Use Disorder; Vaping | interventions — Electronic Nicotine Delivery Systems; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electronic Cigarettes (Active Comparator): Participants in this arm are randomized to receive electronic cigarettes for the 6-week study period.
  Interventions: Drug: Electronic Cigarette
- Nicotine Lozenges (Active Comparator): Participants in this arm are randomized to receive nicotine lozenge for the 6-week study period.
  Interventions: Drug: Nicotine Lozenge

INTERVENTIONS:
Drug: Electronic Cigarette — Electronic Cigarettes are provided to replace tobacco cigarettes
  Arms: Electronic Cigarettes
Drug: Nicotine Lozenge — Nicotine Lozenges are provided to replace tobacco cigarettes
  Arms: Nicotine Lozenges

SUMMARY:
Participants in this randomized clinical trial will be methadone-maintained smokers interested in switching to electronic cigarettes (ECs). There will be a total of 7 study visits over the course of 6 weeks; each visit includes psychometric assessment and biomarker measurements. After completion of the baseline visit, participants will be randomized to either: 1) 6 weeks of EC use (JUUL 5% nicotine pods) or 2) 6 weeks of nicotine replacement therapy (NRT) in the form of nicotine lozenges. EC and NRT use will begin the day after the baseline assessment.

DETAILED DESCRIPTION:
Participants in this randomized clinical trial will be methadone-maintained smokers interested in switching to electronic cigarettes (ECs). There will be a total of 7 study visits over the course of 6 weeks: baseline, 5 weekly check-in (CI) visits, and a 6-week assessment. Baseline assessments will include biomarker measurement, carbon monoxide (CO) readings, smoking history and current cigarette use, spirometry, respiratory symptoms, and tobacco demand. After completion of the baseline visit, participants will be randomized to either: 1) 6 weeks of EC use (JUUL 5% nicotine pods) or 2) 6 weeks of nicotine replacement therapy (NRT) in the form of nicotine lozenges. EC and NRT use will begin the day after the baseline assessment.

All participants will attend weekly brief assessment check-in visits where distribution of either EC or NRT will occur. Check-in assessments will include cigarette use, EC use, NRT use, CO readings, respiratory symptoms, and tobacco demand. At the 6-week assessment, baseline measurements will be repeated to determine changes in the health effects, biomarkers, and combustible cigarette use associated with 6 weeks of EC use, relative to NRT.

This study will be the first to test the potential behavioral and health effects of ECs in smokers with opioid use disorder, a population that is highly dependent on nicotine, highly vulnerable to smoking-related morbidity and mortality, and searching for novel methods to lower smoking-related risks.

ELIGIBILITY:
Inclusion Criteria:

* moderate to heavy cigarette smokers (10 cigarettes/day for > 1 yr; breath CO > 10 ppm)
* have been receiving methadone for at least three months
* attend at least weekly to receive methadone dose
* speak English
* have a telephone or access to a telephone
* are available over the next 6 weeks
* are interested in switching to either electronic cigarettes or nicotine replacement therapy

Exclusion Criteria:

* use of ECs on > 2 of the past 30 days
* currently use medications that may reduce smoking (e.g., bupropion, varenicline, NRT)
* have unstable psychiatric conditions
* have near-daily or daily use of marijuana
* are pregnant
* had a cardiovascular event in the last month
* daily medication for asthma or COPD

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Nicotine Exposure | 6 weeks
  Extent of Nicotine Exposure as measured by urine-based tobacco toxicology assessment at baseline and again at 6-weeks.
FVC Lung Functioning | 6 weeks
  Changes in Forced Vital Capacity (FVC), as measured by spirometry at baseline and again at 6-weeks.
FEV1 Lung Functioning | 6 weeks
  Changes in Forced Expiratory Volume (FEV - during the first second), as measured by spirometry at baseline and again at 6-weeks.
FEV1/FVC Ratio Lung Functioning | 6 weeks
  Changes in FEV1/FVC ratio, as measured by spirometry at baseline and again at 6-weeks.
Smoking Behavior and Experiences | 6 weeks
  Changes in smoking behavior and experiences, as measured by self-report at baseline and again at 6-weeks.
Nicotine Exposure for Complete Switchers | 6 weeks
  Extent of Nicotine Exposure as measured by urine-based tobacco toxicology assessment at baseline and again at 6-week among complete switchers, irrespective of condition, (i.e., exclusive EC/NRT users based on 7-day carbon monoxide (CO)-verified reports at the 6-week time point) relative to dual users and exclusive CC users.
FVC Lung Functioning for Complete Switchers | 6 weeks
  Changes in Forced Vital Capacity (FVC), as measured by spirometry at baseline and again at 6-weeks, among complete switchers, irrespective of condition, (i.e., exclusive EC/NRT users based on 7-day carbon monoxide (CO)-verified reports at the 6-week time point) relative to dual users and exclusive CC users.
FEV1 Lung Functioning for Complete Switchers | 6 weeks
  Changes in Forced Expiratory Volume (FEV - during the first second), as measured by spirometry at baseline and again at 6-weeks, among complete switchers, irrespective of condition, (i.e., exclusive EC/NRT users based on 7-day carbon monoxide (CO)-verified reports at the 6-week time point) relative to dual users and exclusive CC users.
FEV1/FVC Ratio Lung Functioning for Complete Switchers | 6 weeks
  Changes in FEV1/FVC ratio, as measured by spirometry at baseline and again at 6-weeks, among complete switchers, irrespective of condition, (i.e., exclusive EC/NRT users based on 7-day carbon monoxide (CO)-verified reports at the 6-week time point) relative to dual users and exclusive CC users.
Smoking Behavior and Experiences for Complete Switchers | 6 weeks
  Changes in smoking behavior and experiences, as measured by self-report at baseline and again at 6-weeks, among complete switchers, irrespective of condition, (i.e., exclusive EC/NRT users based on 7-day carbon monoxide (CO)-verified reports at the 6-week time point) relative to dual users and exclusive CC users.

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No